CLINICAL TRIAL: NCT06260345
Title: Observatory of Pediatric Severe Communautary Bacterial Infections
Brief Title: CommunautAry Pediatric bacteRial Infection in Intensive CarE Unit
Acronym: CAPRICE
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: GFRUP (Groupe Francophone de Réanimation et d'Urgences Pédiatrique) (Unknown); Groupe de Pathologies Infectieuses Pédiatriques (GPIP) (Other); Centre National de Référence des Streptocoques (Unknown); Centre National de Référence des Pneumocoques (Unknown); Centre National de Référence des Méningocoques et Haemophilus influenzae (Unknown); Centre National de Référence des staphylocoques (Unknown); Centre National de Référence des E. Coli (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAPRICE
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Hospitalized Children; Severe Infection; Invasive Bacterial Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples (blood, pleura, trachea, skine, urine, cerebrospinal fluid etc...) taken during routine care are stored and analysed later for strain characterization by several national reference centers, including those for streptococci, staphylococci, pneumococci, meningococci, hemophilus and Escherichia Coli.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe bacterial infections are a worldwide scourge. However, the epidemiology of this type of infection varies over time. It is therefore essential to monitor them in order to prevent them more effectively. At this time, in France, no monitoring exists for this kind of infections.

DETAILED DESCRIPTION:
The main aim of this study is to assess the number of cases and describe the clinical, biological and microbiological characteristics of these cases of severe communautary invasive bacterial infections in children hospitalized in pediatric intensive care units. In addition, the management of these hospitalized children will be described.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years (only hospitalized children)
* Severe communautary bacterial infection defined by hospitalization in a pediatric intensive care unit (documentation of infection by identification of the bacteria in a sterile environment).

Exclusion Criteria:

* Refusal by one of the parents or by Child in understanding age
* Nosocomial infection

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 ages, with severe communautary invasive bacterial infections, hospitalized in pediatric intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
number of pediatrics cases of severe communautary bacterial infections | 1 year
  Proportion of hospitalized children in intensive care unit due to severe communautary bacterial infections
medical characterisation of children hospitalized for severe communautary bacterial infection case | 1 year
  Assessment of clinical, biological and microbiological characteristics of hospitalized children in intensive care unit due to severe communautary bacterial infections cases

SECONDARY OUTCOMES:
Identify risk factors of serious infection | 1 year
  Describe what is responsible of serious infection
Identify predictive signs of severe cases in infected children. | 1 year
  what are the warning signs of a serious infection?
healthcare used for infected children | 1 year
  Describe healthcare provided during hospitalisation of infected children in order to manage this type of infection
Type of complications | 1 year
  Describe any complications due to infection
Patients outcome | 1 year
  Proportion of patients recovered
treatment used during hospitalisation | 1 year
  type of treatment used during hospitalisation to manage the infection
Bacterial strain characterization | 1 year
  What bacterial strain is involved in the infection?

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, Principal Investigator — CHU Robert Debré, Paris; Corinne Levy, Study Director — Association Clinique Thérapeutique Infantile du val de Marne
Locations (1):
- Association Clinique Thérapeutique Infantile du val de Marne, Créteil, France